CLINICAL TRIAL: NCT03823807
Title: A Multicenter, Open-label, Phase II Study to Evaluate the Safety and Efficacy of SH-1028 in Locally Advanced or Metastatic NSCLC
Brief Title: A Study to Evaluate the Safety and Efficacy of SH-1028 in Locally Advanced or Metastatic NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC013-II-01
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SH-1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH-1028 (Experimental): QD,Oral
  Interventions: Drug: SH-1028

INTERVENTIONS:
Drug: SH-1028 — Oral,100mg or 200mg ,QD, fasted

SUMMARY:
A Phase II, Open Label, Single-arm Study to Assess the Safety and Efficacy of SH-1028 with Locally Advanced/Metastatic Non-Small Cell Lung Cancer whose Disease has Progressed with Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and whose Tumours harbour a T790M mutation within the Epidermal Growth Factor Receptor Gene.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase II study to evaluate the safety and efficacy of SH-1028 in locally advanced or metastatic NSCLC.The trail is divided into two parts:part A is dose extension phase,and Part B is expand sample size phase to confirm the efficacy of SH-1028.Patients must agree to provide a biopsy for central confirmation of T790M mutation status following confirmed disease progression on the most recent treatment regimen. The primary objective of the study is to assess the efficacy of SH-1028 by assessment of Objective Response Rate according to RECIST 1.1 by an Independent Central Review.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, both sexes.
* Histological or cytological confirmation of metastatic or locally advanced, relapsed NSCLC that are not candidates for curative treatment.
* Confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR-TKI sensitivity (including exon 19 deletion, L858R, L861Q, G719X or dual mutation) for treatment-naive NSCLC patients (without systemic therapy or with relapse after previous surgery; patients with locally treatment for non-target lesions are accepted ).(This criteria applies to treatment-naïve NSCLC patients in Part B).
* Patients must have confirmation of T790M+ mutation status, which have experienced disease progression while on a previous continuous treatment with an EGFR-TKI or clinical benefit from EGFR-TKI according to the Jackman criteria while on continuous treatment with an EGFR-TKI (PR/CR, or SD continued ≥6 months); Patients can receive more than one line of systemic therapy. (This criteria applies to EGFR-T790M+ patients in Part A and Part B).
* ECOG score of 0-2 with a minimum life expectancy of 3 months.
* At least 1 lesion that has not previously been irradiated, that can be accurately measured at Baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), which is suitable for accurately repeated measurements.
* Adequate bone marrow reserve or organ function as demonstrated by the following laboratory values: a) absolute neutrophil count ≥ 1.5×109/L; b) platelet count ≥ 100×109/L; c) hemoglobin ≥ 90 g/L; d) ALT ≤ 2.5×ULN if no demonstrable liver metastases, or ALT ≤ 5×ULN in the presence of liver metastases; e) AST ≤ 2.5×ULN if no demonstrable liver metastases, or AST ≤ 5×ULN in the presence of liver metastases; f) Total bilirubin ≤ 1.5×ULN if no liver metastases or ≤ 3×ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases; g) Creatinine ≤ 1.5×ULN, or Creatinine > 1.5×ULN concurrent with creatinine clearance ≥ 50 ml/min (measured or calculated by the Cockcroft- Gault equation).
* Females of child-bearing potential should be using adequate contraceptive measures throughout the study, should not be breast feeding during the study and until 6 months after completion of study, and must have a negative pregnancy test prior to start of dosing.
* Male patients should be willing to use barrier contraception during the study and until 6 months after completion of study (i.e., condoms).
* Do not anticipate other clinical trial in 1 month.
* Patients must sign and date written informed consent prior to admission to the study.

Exclusion Criteria:

* EGFR-TKI treatment within 8 days or approximately 5 times the half-life of the specific drug, whichever is longer, of the first dose study.
* Any cytotoxic chemotherapy or immunological therapy used for a previous treatment regimen or clinical study within 21 days of the first dose of study treatment; Any target therapy(except EGFR-TKIs)and endocrine therapy used for a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
* Ever used the third generation EGFR-TKI, such as Osimertinib, CO-1686, Avitinib, AST2818, HS-10296.
* Major surgery within 4 weeks of the first dose of study treatment.
* Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment.
* The patient is currently using (or cannot discontinue at least 1 week before the first dose of study treatment) a drug or herbal supplement known as a potent inhibitor or inducer of CYP3A4.
* Use large doses of glucocorticoids (eg, >10 mg/day prednisone ) or other immunosuppressive agents within 4 weeks.
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE), Grade 1, at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
* Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids , anticonvulsants and mannitol for at least 4 weeks prior to start of study treatment.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial.
* Active infection (e.g., hepatitis B, hepatitis C or human immunodeficiency virus [HIV]). (HBsAg is positive but HBV-DNA < ULN ,and HCVAb is positive but HCV-RNA<ULN can be accepted.）.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the Screening clinic ECG machine and Fridericia's formula for QT interval correction.
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec).
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Have any other malignant tumor within five years (except clinically cured cervical carcinoma in situ, basal cells or squamous epithelial skin cancer).
* Any seriously abnormal gastrointestinal function would affect uptake, transport and absorption of the drug, such as inability to swallow the study medication, refractory nausea and vomiting, previous significant bowel resection, Recurrent diarrhea, atrophic gastritis (age < 60 years), unhealed serious gastric diseases, Crohn's disease or ulcerative colitis.
* History of hypersensitivity to any active or inactive ingredient of SH-1028 or to a drug with a similar chemical structure or class to SH-1028.
* Women who are breast feeding.
* Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Every 2 cycles (21 days for 1 cycle) until end of treatment, an average of 1 year.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From Baseline up to 30 days after the last dose, an average of 1 year.
Maximum Plasma Concentration (Cmax） | Part A: Day 1 of Cycle 1 and 2 (21 days for 1 cycle).
Area Under the Curve [AUC] | Part A: Day 1 of Cycle 1 and 2 (21 days for 1 cycle).
Progression-free survival (PFS) | Every 2 cycles (21 days for 1 cycle) until end of follow-up, an average of 1 year.
Duration of Response(DOR) | Every 2 cycles (21 days for 1 cycle) until end of treatment, an average of 1 year.
Disease Control Rates(DCR) | Every 2 cycles (21 days for 1 cycle) until end of treatment, an average of 1 year.
Overall survival(OS) | Every 2 cycles (21 days for 1 cycle) until end of treatment; Every 12 weeks until end of follow-up, an average of 2 years.

OTHER OUTCOMES:
Biomakers (eg. AF value of KRAS，MET mutation or other gene mutations ) of drug-resistance measured by next-generation sequencing (NGS). | at end of treatment，an average of 1 years.
  optional，use NGS to analyse the gene associated with NSCLC and to determine the reason of SH-1028-resistance.
Minimum Plasma Concentration (Cmin） | Before administration in Day 1 of cycle 2, 3 and 5 (21 days for 1 cycle).

IPD SHARING:
Plan to Share IPD: No